CLINICAL TRIAL: NCT04988932
Title: Inhalative Stickstoffmonoxid (NO) Behandlung Bei Patienten Mit Schwerem, therapierefraktärem Zerebralen Vasospasmus Nach Subarachnoidalblutung
Brief Title: Inhaled Nitric Oxide Treatment for Aneurysmal SAH Patients With Intractable Cerebral Vasospasm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 019/10
Record Dates: First submitted 2021-07-12; First posted 2021-08-04 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: SAH; Inhaled Nitric Oxide; Cerebral Ischemia; Vasospasm
MeSH Terms: conditions — Brain Ischemia

STUDY DESIGN:
Intervention Model Description: Administration of iNO in SAH patients with severe vasospasm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Administration of iNO in SAH patients with severe vasospasm (Experimental): iNO is started at a dose of 1 parts per million (ppm) and increased stepwise to 2 ppm, 5 ppm, 12 ppm, 25 ppm, until a maximum dose of 40 ppm is reached.
  Interventions: Drug: Inhaled nitric oxide

INTERVENTIONS:
Drug: Inhaled nitric oxide — Each increase of iNO dose is followed by a 10-minute monitoring period and a DSA examination. After reaching the highest effective dose of iNO or the maximum of 40 ppm another DSA is performed. iNO is going to be continued until normalisation of CVS or for a maximum period of 5 days. During iNO treatment a DSA will be performed every 24 hours, followed by a decrease of iNO to the next-lower level. If tapering the iNO concentration is associated with increasing vasospasm, iNO is going to be increased again to the last effective dosage. For cessation of iNO administration, dosage will be tapered every 30 minutes using the same dosage steps as for initiation of iNO treatment. If the duration of iNO treatment will be more than 32 hours, tapering intervals are prolonged to 4 hours. Cessation of iNO will be followed by a DSA.

SUMMARY:
Aneurysmal subarachnoid haemorrhage (aSAH) is a rare but severe subtype of stroke with high mortality and morbidity. Besides rebleeding, delayed cerebral ischaemia and cerebral vasospasm (CVS) are thought to be major reasons for the poor outcome in survivors of aSAH. Despite advances in the detection and treatment of CVS 20-40% of CVS patients experience cerebral Ischaemia. Experimental animal studies for ischaemic stroke, traumatic brain injury, and SAH showed that inhaled nitric oxide (iNO) selectively dilates cerebral arteries and arterioles in hypoperfused brain tissue. The investigators therefore performed this prospective pilot study to evaluate the effects of iNO on cerebral perfusion in patients with refractory vasospasm after aSAH.

DETAILED DESCRIPTION:
Aneurysmal subarachnoid haemorrhage (aSAH) is a rare but severe subtype of stroke with high mortality and morbidity. Besides rebleeding, delayed cerebral ischaemia and cerebral vasospasm (CVS) are thought to be major reasons for the poor outcome in survivors of aSAH. CVS, thought to be caused by blood breakdown products, peak in the second week after hemorrhage and affect up 88% of patients with severe aSAH. Despite advances in the detection and treatment of CVS there is no established therapy and up 40% of patients experience cerebral ischemia. In symptomatic vasospasm and cerebral hypoperfusion various treatments like induced hypertension, angioplasty and intraarterial vasodilators are used as rescue therapies. Yet, their effect is not proven.

In recent experimental studies, inhaled nitric oxide (iNO) has been shown to induce a selective dilation of cerebral arteries and arterioles in hypoperfused brain tissue [8, 9]. After experimental SAH in mice, iNO significantly reduced the number and severity of SAH-induced spasms of cerebral microvessels, thereby improving cerebral perfusion. Inhaled NO has regulatory approval in man by the Food and Drug Administration (FDA) and by the European Medicines Agency (EMA) for the treatment of several pulmonary pathologies. At first the efficacy of iNO was thought to be limited to the lungs but, based on the results of the experimental studies the investigators hypothesised that iNO may relieve CVS and improve cerebral perfusion in patients with aSAH.

The investigators performed this prospective trial to evaluate the effect of iNO on cerebral perfusion in patients with severe refractory CVS. Only patients with refractory CVS after maximum conservative treatment were included. Inhaled NO was administered to a maximum dose of 40ppm. The effect was assessed by digital subtraction angiography (DSA), tissue oxygen partial pressure (PtiO2), transcranial Doppler (TCD), and CT perfusion (CTP) imaging. Patiente outcome is assessed at 12 weeks an 6 months after hemorrhage and included NIHSS, Mini Mental State (MMS) test, and modified Rankin Scale (mRS).

ELIGIBILITY:
Inclusion Criteria:

* aSAH of all severities
* Aneurysm treated by either surgical clipping or endovascular coiling
* Age between 18 - 80 years
* Proven CVS
* Cerebral hypoperfusion and neurological deficit despite treatment (oral nimodipine, induced hypertension, hypervolaemia, central venous pressure > 6 mmHg)
* A negative pregnancy test in women
* Signed informed consent from the next of kin and an independent physician

Exclusion Criteria:

* Unsecured aneurysm
* Cerebral infarction on imaging in the downstream brain parenchyma of spastic vessel
* Cerebral herniation
* Intracranial pressure > 25 mmHg
* Pregnancy
* Mean arterial pressure ≤ 90 mmHg despite catecholamines

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-07-31 (Actual); Primary Completion 2019-07-28 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Improvement of severe vasospasm in digital subtraction angiography | Up to 5 days
  > 10% increase in diameter of the vasospastic target vessel compared to baseline
Improvement of severe vasospasm in tissue oxygen partial pressure (PtiO2) | Up to 5 days
  An increase of more than 5 mmHg with constant fraction of inspired oxygen (FiO2)
Improvement of severe vasospasm in transcranial Doppler | Up to 5 days
  A decrease of more than 30 cm/s
Improvement of severe vasospasm in CT perfusion | Day 2
  A reduction in the number of Region of interest with impaired perfusion (MTT > 6·5 s)

SECONDARY OUTCOMES:
Intracranial pressure | Up to 5 days
  Intracranial pressure using an external ventricular drain catheter
Assessment of ischaemic events by CT Scan | 12 weeks after SAH

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Beck, MD, Principal Investigator — Inselspital Bern, Department of Neurosurgery
Locations (1):
- Department of Neurosurgery, University Hospital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Terpolilli NA, Feiler S, Dienel A, Muller F, Heumos N, Friedrich B, Stover J, Thal S, Scholler K, Plesnila N. Nitric oxide inhalation reduces brain damage, prevents mortality, and improves neurological outcome after subarachnoid hemorrhage by resolving early pial microvasospasms. J Cereb Blood Flow Metab. 2016 Dec;36(12):2096-2107. doi: 10.1177/0271678X15605848. Epub 2015 Nov 2. PMID 26661144
- [Background] Terpolilli NA, Kim SW, Thal SC, Kataoka H, Zeisig V, Nitzsche B, Klaesner B, Zhu C, Schwarzmaier S, Meissner L, Mamrak U, Engel DC, Drzezga A, Patel RP, Blomgren K, Barthel H, Boltze J, Kuebler WM, Plesnila N. Inhalation of nitric oxide prevents ischemic brain damage in experimental stroke by selective dilatation of collateral arterioles. Circ Res. 2012 Mar 2;110(5):727-38. doi: 10.1161/CIRCRESAHA.111.253419. Epub 2011 Dec 29. PMID 22207711
- [Background] Terpolilli NA, Brem C, Buhler D, Plesnila N. Are We Barking Up the Wrong Vessels? Cerebral Microcirculation After Subarachnoid Hemorrhage. Stroke. 2015 Oct;46(10):3014-9. doi: 10.1161/STROKEAHA.115.006353. Epub 2015 Jul 7. No abstract available. PMID 26152299
- [Background] Terpolilli NA, Kim SW, Thal SC, Kuebler WM, Plesnila N. Inhaled nitric oxide reduces secondary brain damage after traumatic brain injury in mice. J Cereb Blood Flow Metab. 2013 Feb;33(2):311-8. doi: 10.1038/jcbfm.2012.176. Epub 2012 Nov 28. PMID 23188422
- [Background] Germann P, Braschi A, Della Rocca G, Dinh-Xuan AT, Falke K, Frostell C, Gustafsson LE, Herve P, Jolliet P, Kaisers U, Litvan H, Macrae DJ, Maggiorini M, Marczin N, Mueller B, Payen D, Ranucci M, Schranz D, Zimmermann R, Ullrich R. Inhaled nitric oxide therapy in adults: European expert recommendations. Intensive Care Med. 2005 Aug;31(8):1029-41. doi: 10.1007/s00134-005-2675-4. Epub 2005 Jun 23. PMID 15973521
- [Background] Griffiths MJ, Evans TW. Inhaled nitric oxide therapy in adults. N Engl J Med. 2005 Dec 22;353(25):2683-95. doi: 10.1056/NEJMra051884. No abstract available. PMID 16371634